CLINICAL TRIAL: NCT01003327
Title: Comparison of the I-gel Laryngeal Mask and the Classic Laryngeal Mask in Patients With a BMI>25 During Elective Surgery
Brief Title: Comparison of the I-gel Laryngeal Mask and the Classic Laryngeal Mask in Patients With a BMI>25
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Dr. Ulrike Weber, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 354/2009
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2009-10

CONDITIONS: Surgery; Intubation
Keywords: laryngeal mask, leak pressure; leak pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- I-gel inserted first (Other): The I-gel airway is insewrted first, then the LMA-Unique
  Interventions: Device: I-gel
- LMA-Unique inserted first (Other): LMA-Unique airway is inserted first, then the I-gel
  Interventions: Device: LMA-Unique

INTERVENTIONS:
Device: I-gel — intubation with I-gel airway
  Arms: I-gel inserted first
Device: LMA-Unique — LMA-Unique airway is inserted first, then the I-gel
  Arms: LMA-Unique inserted first

SUMMARY:
The intention of this study is to compare the performance of the single-use I-gel laryngeal mask with the classic laryngeal mask in 50 patients with a BMI>25 during elective surgery. Primary outcome is the leak pressure. Secondary outcomes include ease and duration of insertion.

DETAILED DESCRIPTION:
Inclusion criteria of this randomized cross-over study are: BMI > 25, elective surgery in supine position, age>18 years, ASA I-II; Exclusion criteria are: difficult airway, pregnancy, history of reflux or gastrointestinal disorders, abdominal or thoracic surgery; In this cross-over trial both airway devices are inserted in the same patient, the order of insertion is randomized. Patient receive monitoring with blood pressure, ECG and pulse oxymetry during operation. Anaesthesia is induced intravenously using fentanyl (0.001 mg/kg) and propofol (3-5 mg/kg). The I-gel laryngeal mask is inserted with a gastric tube. The classic laryngeal mask was cuffed after insertion with a cuff pressure of 60 cmH2O. The first device is removed 5 minutes after insertion and replaced by the second device. Ease of insertion is graded as very easy=1, easy=2, difficult=3 and very difficult=4. Leak pressure is measured by two tests: In the first test the spill valve is closed at a fresh gas flow of 6l/min and the minimum airway pressure at which gas leaked around the airway device is recorded by listening for an audible leak. In the second test leakage is measured during pressure controlled ventilation. Therefore we administer a fresh gas flow of 3l/min, FiO2 of 50%, inspiration to expiration ratio of 1:2 and a frequency of breathing of 12. Leakage can be measured by the respirator. We record inspiration pressure, mean pressure, plateau pressure, tidal volume and peep at which the first measurable leakage occurred.

For statistical analysis we will use t-tests with a power of 80% and a p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 25, elective surgery in supine position,
* age > 18 years,
* ASA I-II;

Exclusion Criteria:

* difficult airway, pregnancy,
* history of reflux or gastrointestinal disorders,
* abdominal or thoracic surgery;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
leak pressure of the laryngeal masks | directly after insertion of the laryngeal mask

SECONDARY OUTCOMES:
Insertion time and ease of insertion of the laryngeal mask | during insertion of the laryngeal mask

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Weber, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical university of vienna, General hospital of Vienna, Vienna, Vienna, Austria